CLINICAL TRIAL: NCT02446496
Title: Comparative Randomized, Single Dose, Two-way Crossover, Open-label Study to Determine the Bioequivalence of Cefadroxil From Duricef 1 gm Film Coated Tablets (Smithkline Beecham Egypt, LLC Affiliated Co. to GalaxoSmithKline ) and Biodroxil 1 gm Film Coated Tablets (Kahira Pharm &Chem .Ind. Co. for Novartis Pharma ) After a Single Oral Dose Administration of Each to Healthy Adults Under Fasting Conditions
Brief Title: A Bioequivalence Study of Cefadroxil Film Coated Tablets After A Single Oral Dose Administration to Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 201529
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Infections, Urinary Tract
Keywords: Bioequivalence; film coated tablets; cefadroxil
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cefadroxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Subjects will receive a single oral dose of cefadroxil tablet manufactured by GSK under fasting condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of cefadroxil tablet manufactured by NP under fasting condition in treatment period 2
  Interventions: Drug: Cefadroxil tablets manufactured by GSK; Drug: Cefadroxil tablets manufactured by NP
- Group B (Experimental): Subjects will receive a single oral dose of cefadroxil tablet manufactured by NP under fasting condition in treatment period 1 followed by 7 days washout interval from the first study drug administration. After the washout interval the subjects will receive a single dose of cefadroxil tablet manufactured by GSK under fasting condition in treatment period 2
  Interventions: Drug: Cefadroxil tablets manufactured by GSK; Drug: Cefadroxil tablets manufactured by NP

INTERVENTIONS:
Drug: Cefadroxil tablets manufactured by GSK — Cefadroxil tablets manufactured by GSK contains 1 mg of Cefadroxil
Drug: Cefadroxil tablets manufactured by NP — Cefadroxil tablets manufactured by NP contains 1 mg of Cefadroxil

SUMMARY:
This is an open-label, randomized, single dose, two-sequence two-period crossover study, separated by 7 days washout interval from the first Study Drug Administration. This study is conducted to determine the bioequivalence of cefadroxil from DURICEF™ film coated tablets manufactured by Smithkline Beecham Egypt, LLC affiliated co. to GalaxoSmithKline (GSK) and cefadroxil from BIODROXIL™ film coated tablets manufactured by Kahira Pharm &Chem .Ind. Co . for Novartis Pharma (NP) after a single oral dose administration of each to healthy adult subjects under fasting conditions. In Period 1, subjects will be randomized to receive cefadroxil tablet manufactured by either GSK or NP. Following a washout of at least 7 days, subjects will be crossed over in Period 2 to receive the cefadroxil tablet that they did not receive in Period 1. DURICEF is a trademark of the GSK group of companies. BIODROXIL is a trademark of Sandoz.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, age 18 to 55 years, inclusive.
* Body weight within 15 percent of normal range according to the accepted normal values for body mass index (BMI).
* Medical demographics without evidence of clinically significant deviation from normal medical condition.
* Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.
* Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

* Subjects with known allergy to the products tested.
* Subjects whose values of BMI were outside the accepted normal ranges.
* Female subjects who were pregnant, nursing or taking birth control pills.
* Medical demographics with evidence of clinically significant deviation from normal medical condition.
* Results of laboratory tests which are clinically significant.
* Acute infection within one week preceding first study drug administration.
* History of drug or alcohol abuse.
* Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.
* Subject is on a special diet (for example subject is vegetarian).
* Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.
* Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.
* Subject has a history of severe diseases which have direct impact on the study.
* Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.
* Subject intends to be hospitalized within 6 weeks after first study drug administration.
* Subjects who, through completion of this study, would have donated more than 500 milliliter (mL) of blood in 7 days, or 750 mL of blood in 30 days, 1000 mL in 90 days, 1250 mL in 120 days, 1500 mL in 180 days, 2000 mL in 270 days, 2500 mL of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2014-04-08 (Actual); Study Completion 2014-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 201529 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 24 participants were enrolled in from March-2014 to April-2014. During each study period participants received test (treatment A-cefadroxil tablet) and reference (treatment B-cefadroxil tablet) products.
Pre-assignment Details: Total of 28 participants were screened, out of which 4 were screen failure. Of 4 participants, 1 withdrawn due to significant variation in laboratory results and 3 withdrawn upon their will.
Groups:
- Treatment A-cefadroxil 1 gm + Treatment B-cefadroxil 1 gm: In each period of the study, participants received one tablet of treatment A (cefadroxil 1 gram [gm] film coated [F.C.] tablet) or treatment B (cefadroxil 1 gm F.C. tablet), given with 240 ml water. Water was at room temperature and measured with a 250 ml cylinder according to a plan of randomization. The study drug administration took place between 09:00 ante meridiem (am) and 09:46 am for both periods in the morning of study Day 1 of each study period. A washout period of 7 days between the two study drug administrations was allowed.
Period: Overall Study
Arm/Group | Treatment A-cefadroxil 1 gm + Treatment B-cefadroxil 1 gm
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment A-cefadroxil 1 gm + Treatment B-cefadroxil 1 gm
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.46 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  Oriental | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximal Measured Plasma Concentration (Cmax) After a Single Dose
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at indicated time points of each treatment period. Cmax was defined as maximal measured plasma concentration over the time span specified.
Time Frame: Pre-dose (0.00) and 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 4.00, 6.00, 8.00, 10.00 and 12.00 hours post-dose in each treatment period.
Population: All subject population: who were crossed over and completed the balance design, were included in the calculation. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Groups:
- Treatment A-cefadroxil 1 gm: In each period of the study, participants received one tablet of treatment A (cefadroxil 1 gm F.C. tablet), given with 240 ml water. Water was at room temperature and measured with a 250 ml cylinder according to a plan of randomization. The study drug administration took place between 09:00 am and 09:46 am for both periods in the morning of study Day 1 of each study period. A washout period of 7 days between the two study drug administrations was allowed.
- Treatment B-cefadroxil 1 gm: In each period of the study, participants received one tablet of treatment B (cefadroxil 1 gm F.C. tablet), given with 240 ml water. Water was at room temperature and measured with a 250 ml cylinder according to a plan of randomization. The study drug administration took place between 09:00 am and 09:46 am for both periods in the morning of study Day 1 of each study period. A washout period of 7 days between the two study drug administrations was allowed.
Arm/Group | Treatment A-cefadroxil 1 gm | Treatment B-cefadroxil 1 gm
Number analyzed (Participants) | 24 | 24
Microgram per milliliter | 28.18 (8.12) | 29.20 (8.80)
Statistical Analysis 1: Comparison: Treatment A-cefadroxil 1 gm vs Treatment B-cefadroxil 1 gm; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; Point estimate percent = 95.91, 90% CI 2-sided [85.67 to 107.37]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) and Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-infinity)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. Area under the plasma concentration-time curve from time zero (0) to the last measurable concentration (t), as calculated by the linear trapezoidal method. Area under the plasma concentration-time curve from time zero (0) to infinity (AUC0-infinity) was calculated as the sum of the AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant (Ke), where first-order elimination or terminal rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram.hour per milliliter
Arm/Group | Treatment A-cefadroxil 1 gm | Treatment B-cefadroxil 1 gm
Number analyzed (Participants) | 24 | 24
Microgram.hour per milliliter
  AUC(0-t) | 106.55 (28.64) | 102.21 (26.06)
  AUC(0-infinity) | 111.71 (30.15) | 106.08 (26.40)
Statistical Analysis 1: Comparison: Treatment A-cefadroxil 1 gm vs Treatment B-cefadroxil 1 gm; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; Point estimate percent = 102.31, 90% CI 2-sided [90.46 to 115.70] — Comparison of AUC (0-t) between Treatment A and Treatment B
Statistical Analysis 2: Comparison: Treatment A-cefadroxil 1 gm vs Treatment B-cefadroxil 1 gm; Test type: Non-Inferiority or Equivalence — Bioequivalence is established when 90% Confidence Interval falls within 80-125%; Point estimate percent = 103.13, 90% CI 2-sided [91.19 to 116.62] — Comparison of AUC(0-infinity) between Treatment A and Treatment B

3. Secondary Outcome: Time of the Maximum Plasma Concentration (T-max) and Terminal Half- Life (T-half)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. If the maximum value occurs at more than one point T-max was defined as the first time point with this value. The elimination or terminal half-life was calculated by dividing 0.693 (natural logarithm of 2) with lambda z, where lambda z is the terminal phase rate constant estimated by linear regression analysis of the log transformed concentration-time data after each single dose.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A-cefadroxil 1 gm | Treatment B-cefadroxil 1 gm
Number analyzed (Participants) | 24 | 24
Hour
  T-max | 1.50 [0.75 to 4.00] | 1.50 [0.75 to 3.00]
  T-half | 2.28 [1.89 to 3.13] | 2.10 [1.72 to 3.85]
Statistical Analysis 1: Comparison: Treatment A-cefadroxil 1 gm vs Treatment B-cefadroxil 1 gm; Test type: Superiority or Other; p = 0.2670, Wilcoxon's Signed-Rank Test; Comparison of T-max between Treatment A and Treatment B

4. Secondary Outcome: Apparent First-order Elimination or Terminal Rate Constant (Ke)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. Apparent first-order elimination or terminal rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: All subject population. All participants were present at the time of measurement.
Measure: Mean (Standard Deviation); unit: Per hour
Arm/Group | Treatment A-cefadroxil 1 gm | Treatment B-cefadroxil 1 gm
Number analyzed (Participants) | 24 | 24
Per hour | 0.30 (0.03) | 0.33 (0.05)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAE) were reported through out the study (up to 11 days)
Description: An AE and SAE were reported in all subject population.
Arm/Group | Treatment A-cefadroxil 1 gm | Treatment B-cefadroxil 1 gm
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.